CLINICAL TRIAL: NCT03689452
Title: The Effect of Platelet Rich Plasma on Non-scarring Alopecia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Eclipse Aesthetics, LLC (Other)
Responsible Party: Principal Investigator, Hooman Khorasani, Clinical Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 18-1714
Record Dates: First submitted 2018-09-20; First posted 2018-09-28 (Actual); Results first posted 2020-10-30 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Androgenetic Alopecia; Alopecia
MeSH Terms: conditions — Alopecia | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Control (Placebo Comparator): 15 participants will receive 3 mL of preservative free normal saline injected in a standardized pattern with each injection 1-2 cm apart with 0.2 to 0.3 mL per injection. Participants will receive this treatment at weeks 0, 4, 8, and 24.
  Interventions: Drug: Normal saline
- Treatment (Experimental): 15 participants will receive 3-6 mL of platelet rich plasma injected in a standardized pattern with each injection 1-2 cm apart with 0.2 to 0.3 mL per injection. Participants will receive this treatment at weeks 0, 4, 8, and 24.
  Interventions: Device: Platelet Rich Plasma

INTERVENTIONS:
Device: Platelet Rich Plasma — Platelet Rich Plasma (PRP) is defined as an autologous concentration of human platelets that is 3 to 5 times greater than physiologic concentration of platelets in whole blood. Using the Eclipse PRP system, the participants PRP will be attained. The PRP will then be used as described in the arm/group description section.
  Arms: Treatment
Drug: Normal saline — Preservative-free normal saline will be used as described in arm/group description section.
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy of platelet rich plasma (PRP) injections for non-scaring alopecia in women. A randomized, placebo-controlled clinical trial will be performed where patients with non-scarring alopecia will either receive injections of their own PRP or injections of normal saline (placebo). Patients in the treatment group (Group A) will have a small amount of their own blood drawn and have their PRP injected into their scalp four times. The injections will be given at weeks zero, four, eight, and twenty four. The placebo group (Group B) will be given the same schedule but will receive sham injections only and will not have any blood drawn. Both groups will have clinical data collected at all visits, including a screening visit before enrollment and a final assessment visit at week 40, for a total of 6 study visits per patient. Data collection will include representative photographs of the scalp and measurements of hair thickness. The results from the two groups will then be compared.

In summary, all study participants will have a screening visit before enrollment, four study visits for sub-dermal scalp injections, and one final assessment visit at week 40.

ELIGIBILITY:
Inclusion Criteria:

1. Must understand and voluntarily sign an informed consent form
2. Must be female between the ages of 18 and 65 years at the time of consent
3. Must be able to adhere to the study visit schedule and other protocol requirements
4. Documented platelet count above 150,000 platelets per microliter within 6 months prior to enrollment

Exclusion Criteria:

1. Previous or current use in the last 1 year of finasteride, minoxidil topical or oral, or spironolactone
2. A diagnosis of non-androgenic alopecia (i.e: another diagnosis for the alopecia )
3. No Baseline ferritin, thyroid-stimulating hormone, platelet count, and a negative urine pregnancy test in any pre-menopausal female in past 12 months.
4. Active skin disease (Psoriasis or severe seborrheic dermatitis) of the scalp
5. Scalp infection
6. Severe active blood infection
7. Cuts or abrasions on the scalp
8. History of surgical hair restoration
9. Current or recent malignancy
10. History of systemic chemotherapy or radiation
11. History of thyroid dysfunction
12. History of autoimmune disorder (specifically Graves disease, hashimoto thyroiditis, or systemic lupus erythematosus)
13. Tendency to develop keloids
14. Nonsteroidal anti-inflammatory or Vitamin E discontinued in the last 7-14 days
15. Platelet dysfunction syndrome
16. Thrombocytopenia less than 150,000
17. Diagnosis of hypofibrinogenemia
18. Anticipated pregnancy or trying to become pregnant in the next 2 years

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-06-03 (Actual); Study Completion 2019-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hooman Khorasani, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Raw individual participant data will not be shared with other researchers in an effort to preserve participant confidentiality.

RESULTS

PARTICIPANT FLOW:
Groups:
- Platelet Rich Plasma (PRP) Group: 4.0 mL of Platelet Rich Plasma (PRP), an autologous concentration of human platelets that is 3 to 5 times greater than physiologic concentration of platelets in whole blood, injected in a standardized pattern with each injection 1-2 cm apart with 0.2 mL per injection.
- Placebo Group: 4.0 mL of Preservative-free normal saline injected in a standardized pattern with each injection 1-2 cm apart with 0.2 mL per injection.
Period: Overall Study
Arm/Group | Platelet Rich Plasma (PRP) Group | Placebo Group
Started | 15 | 15
Completed | 14 | 14
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Platelet-rich Plasma Group: 4.0 mL of Platelet Rich Plasma (PRP), an autologous concentration of human platelets that is 3 to 5 times greater than physiologic concentration of platelets in whole blood, injected in a standardized pattern with each injection 1-2 cm apart with 0.2 mL per injection.
- Total: Total of all reporting groups
Arm/Group | Platelet-rich Plasma Group | Placebo Group | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Full Range); unit: years] | 47 [28 to 70] | 53 [27 to 85] | 50 [27 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 8 | 7 | 15
  Hispanic | 5 | 7 | 12
  Other | 2 | 1 | 3
Hair Loss [Mean (Full Range); unit: months] | 67 [8 to 204] | 93 [8 to 300] | 80 [8 to 300]
Ludwig Score [Count of Participants; unit: Participants] — I is appreciable thinning of the crown hair, II is increased territorial involvement and scalp visibility, and III is total denudation of the areas involved in I and II
  Participants
    I | 8 | 9 | 17
    II | 6 | 5 | 11
    III | 1 | 1 | 2
Hair Density [Mean (Full Range); unit: hairs/cm^2] | 556 [102 to 830] | 598 [321 to 807] | 577 [102 to 830]
Hair Caliber [Mean (Full Range); unit: mm] | 0.0509 [0.0300 to 0.0690] | 0.0570 [0.0400 to 0.0800] | 0.0540 [0.0300 to 0.0800]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Improvement
Description: Number of participants with improvement by qualitative global assessment of hair growth using photography. Photographs of the scalp with standard digital camera used to assess overall change in hair appearance on a macroscopic level. This will be done using the Ludwig Classification system.
  I is appreciable thinning of the crown hair, II is increased territorial involvement and scalp visibility, and III is total denudation of the areas involved in I and II
Time Frame: through study completion, 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Platelet-rich Plasma Group | Placebo Group
Number analyzed (Participants) | 14 | 14
Participants | 8 | 1

2. Primary Outcome: Change in Hair Caliber Using Trichoscopy
Description: Change in Hair Caliber using trichoscopy as compared to baseline. Trichoscopy is a microscope used to assess hair. This was used to measure hair caliber in millimeters.
Time Frame: Week 8 and 24
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Platelet-rich Plasma Group | Placebo Group
Number analyzed (Participants) | 14 | 14
mm
  Week 8 | 0.0043 (0.0024) | -0.0034 (0.0049)
  Week 24 | 0.0053 (0.0061) | -0.0060 (0.0063)

3. Primary Outcome: Change in Hair Density Using Trichoscopy
Description: Change in Hair Density using trichoscopy as compared to baseline. Trichoscopy is a microscope used to assess hair. This was used to measure hair density (number of hairs in a square centimeter of scalp).
Time Frame: Week 8 and 24
Measure: Mean (Standard Deviation); unit: hairs/cm^2
Arm/Group | Platelet-rich Plasma Group | Placebo Group
Number analyzed (Participants) | 14 | 14
hairs/cm^2
  Week 8 | 71.1 (40.8) | -26.7 (46.7)
  Week 24 | 105.9 (102.9) | -52.4 (53.0)

4. Secondary Outcome: Qualitative Assessment of Hair Growth
Description: Surveys will be distributed to assess participant opinion regarding overall hair growth after treatment. This will be done using a hair growth scale in which 0 is no improvement in hair growth and 10 is greatly improved hair growth.
Time Frame: Week 40
Population: Data not collected
Arm/Group | Platelet-rich Plasma Group | Placebo Group
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Qualitative Assessment of Pain Associated With the Treatment
Description: Surveys will be distributed to assess participant opinion regarding the degree of pain associated with the treatment. This will be done using a pain scale of 0 to 10 with 0 being no pain and 10 being worst pain ever.
Time Frame: Week 40
Population: Data not collected
Arm/Group | Platelet-rich Plasma Group | Placebo Group
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Qualitative Assessment of Adverse Effects Associated With the Treatment
Description: Questionnaires will be distributed to assess participant opinion regarding adverse effects associated with the treatment. This will be assessed via a multiple choice questionnaire with the following options:
  i. Headache ii. Scalp tightness iii. Swelling iv. Redness v. Post-injection bleeding vi. Infection vii. Nerve damage viii. Other: ____________________ ix. None
Time Frame: Week 40
Population: Data not collected at 40 weeks.
Arm/Group | Platelet-rich Plasma Group | Placebo Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Platelet-rich Plasma Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 11/14 | 6/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Platelet-rich Plasma Group (N=14) | Placebo Group (N=14)
Headache (Nervous system disorders) | 7 | 4
Scalp tightness (General disorders) | 7 | 3
Swelling (Skin and subcutaneous tissue disorders) | 4 | 0
Redness (Skin and subcutaneous tissue disorders) | 2 | 0
Post-injection bleeding (Blood and lymphatic system disorders) | 1 | 0
Tingling (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-09-21): https://cdn.clinicaltrials.gov/large-docs/52/NCT03689452/SAP_001.pdf
  • Study Protocol (2018-09-21): https://cdn.clinicaltrials.gov/large-docs/52/NCT03689452/Prot_002.pdf